CLINICAL TRIAL: NCT00850694
Title: Assessment of Prevalence of Vitamin D Deficiency in Obese Adolescent Girls and Influence of Vitamin D on Insulin Secretion and Sensitivity
Brief Title: Vitamin D Deficiency in Obese Adolescent Girls and Influence of Vitamin D on Insulin Secretion and Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ambika Ashraf, M.D., Assistant Professor, Pediatrics, University of Alabama at Birmingham
Other Study IDs: F061228001
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2011-09

CONDITIONS: Vitamin D Deficiency; Obesity; Insulin Resistance
Keywords: Vitamin D deficiency; Obesity; Insulin resistance; Glucose tolerance
MeSH Terms: conditions — Vitamin D Deficiency; Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Obese female adolescents

SUMMARY:
Sub-clinical vitamin D deficiency is a commonly unrecognized disorder in obese adolescents. The investigators hypothesize vitamin D deficiency will be highly prevalent in obese adolescents and those who are vitamin D deficient will be more insulin resistant.

DETAILED DESCRIPTION:
This is a cross-sectional study of obese female adolescents matched for age, sex and pubertal staging. Serum 25-OH vitamin D, intact PTH , lipid profile, serum CRP measurements and oral glucose tolerance tests (with glucose and insulin level measurements) will be done to assess the prevalence of vitamin D deficiency and to assess the insulin sensitivity- resistance indices.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents
* Obese: BMI > 95th percentile
* Menarchal
* Tanner stage ≥ 4

Exclusion Criteria:

* Children with diabetes, other endocrine or acute or chronic medical illnesses, children on oral contraceptive pills, diuretics and anticonvulsant medications

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese female adolescents
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2007-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of subclinical vitamin D deficiency in obese female adolescents. | At study entry

SECONDARY OUTCOMES:
To assess the relationship of serum 25 (OH) D statuses to insulin and glucose concentrations during an OGTT and to serum transaminases and CRP. | At study entry

CONTACTS AND LOCATIONS:
Overall Officials: Ambika Ashraf, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's Hospital, Universiy of Alabama at Birmingham, Birmingham, Alabama, United States